CLINICAL TRIAL: NCT04385030
Title: Transcranial Direct Current Stimulation and Mirror Therapy in Neuropathic Pain
Brief Title: Neurostimulation and Mirror Therapy in Traumatic Brachial Plexus Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Principal Investigator and Professor, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NeuroPain
Record Dates: First submitted 2020-02-23; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Direct Current Stimulation; Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ETCC Active associated with Mirror Therapy (TE) (Active Comparator): The study will consist of 12 sessions, being carried out over a period of 1 month, with 3 weekly sessions on consecutive days, where each patient will receive ETCC for 30 minutes concomitantly with ET. Outcome assessments will be performed before the beginning of the protocol on the base (T0) and immediately after the end of the 12 sessions (T1).
  Interventions: Device: TRANSCRANIAL DIRECT CURRENT STIMULATION AND MIRROR THERAPY
- ETCC simulated associated with Mirror Therapy (TE) (Sham Comparator): The study will consist of 12 sessions, being carried out over a period of 1 month, with 3 weekly sessions on consecutive days, where each patient will receive ETCC for 30 minutes concomitantly with ET. Outcome assessments will be performed before the beginning of the protocol on the base (T0) and immediately after the end of the 12 sessions (T1).
  Interventions: Device: TRANSCRANIAL DIRECT CURRENT STIMULATION AND MIRROR THERAPY

INTERVENTIONS:
Device: TRANSCRANIAL DIRECT CURRENT STIMULATION AND MIRROR THERAPY — The study will consist of 12 sessions, carried out over a period of 1 month, with 3 weekly sessions on consecutive days, where each patient will receive ETCC for 30 minutes concomitantly with ET. Outcome assessments will be performed before the beginning of the protocol on the base (T0) and immediately after the end of the 12 sessions (T1).

SUMMARY:
Traumatic injuries of the brachial plexus cause sufficient weakness to affect the individual in its various aspects, limiting the execution of Activities of Daily Living, leading to highly disabling, and often definitive, clinical conditions with serious socioeconomic consequences. It causes motor, sensory and autonomic deficits, directly compromising the quality of life and functional performance of these individuals. It is a complex condition, whose recovery is usually slow and costly, in addition to often requiring surgery and rehabilitation. Among the therapeutic possibilities, the non-invasive neuromodulation techniques stand out, especially the Transcranial Direct Current Stimulation (ETCC) and the Mirror Therapy (ET). In this context, the present study aims to analyze the effectiveness of the ETCC technique combined with ET in the treatment of patients with pain due to trauma to the brachial plexus, investigating the degree of improvement in pain intensity, functionality, quality of life and mood of these patients, comparing the onset with immediately after applying the techniques.

DETAILED DESCRIPTION:
For this, a pilot clinical trial, placebo-controlled, blind and randomized, will be carried out, involving patients with traumatic brachial plexus injury, submitted to sessions of ETCC and mirror therapy. Participants will be randomly allocated to 1 of 2 groups: the first will receive active ETCC associated with TE and the second will receive simulated ETCC in conjunction with TE. The study will consist of 12 sessions, conducted over a period of 1 month, with 3 sessions weekly on consecutive days, where each patient will receive ETCC for 30 minutes concomitantly with ET. Assessments will be performed before the beginning of the protocol (baseline) and immediately after the end of the 12 sessions. The TCT-Research device, developed by Trans Cranial Technologies Ltda for ETCC and a rectangular platform with the dimensions of 40x70 cm, with a mirror sagittally coupled to the TE will be used. To assess the outcomes, EVA, McGill's Questionnaire, BPI, BDI, IDATE, SF-36 and CIF will be applied. For all analyzes, the statistical software SPSS (SPSS Inc, Chicago IL, USA) for Windows, version 20.0, will be used and considered significant, an alpha value of 5% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Score of 4 to 10 points on the Visual Analogue Scale;
* Persistent pain and refractory to clinical treatment for at least 3 months;
* Appropriate pharmacological treatment for pain for at least 1 month before the start of the study.

Exclusion Criteria:

* Patients with other neurological diseases;
* Past history of substance abuse;
* Contraindications for ETCC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline and after 4 weeks
  Visual analog scale (VAS) - One-dimensional instrument for assessing pain intensity. It is a line with the ends numbered 0-10. At one end line is marked "no pain" and on the other "worse pain imaginable".
Changes in pain interference in activities of daily living | Baseline and after 4 weeks
  1 - Brief Pain Inventory - reduced form (Brief Pain Inventory - BPI): Multidimensional instrument, which makes use of a scale of 0-10 to graduate the following items: intensity, pain interference on ability for walking, daily activities of the patient, at work, social activities, mood and sleep.
Change in pain characteristics | Baseline and after 4 weeks
  2 - McGill Pain Questionnaire - MPQ): The descriptors are divided into four groups: sensory discriminative, motivational affective, cognitive evaluative, and miscellaneous. The numerical index of descriptors is the number of words chosen by the patient to characterize your pain, being at most a word of each subgroup with a maximum value of 20. The pain index is calculated by adding the values of intensity of each descriptor (0-5), having this maximum 78.

SECONDARY OUTCOMES:
Quality of life (SF-36) | Baseline and after 4 weeks
  The Medical Outcomes Short-Form Health Survey (SF-36) - a general health assessment instrument, originally created in English, which is easy to administer and understand. It consists of 36 questions, covering eight components, functional capacity, physical aspects, pain, general health status, vitality, social aspects, emotional aspects and mental health assessed by 35 questions and one more comparative question between current and health one year ago.
Functionality | Baseline and after 4 weeks
  International Classification of Functionality, Disability and Health (ICF) - formed by categories and their subdivisions, or constructs, of different dimensions, including parts of the body. It covers functionality as activity and participation, that is, what human beings can do in different situations or under the influence of different environments, for example. Each category or construct is related to a set that must be completed by qualifiers, numbers that indicate the magnitude of a problem within a specific category. In general, the user must select the categories and qualifiers that identify and express each case.11 The classification must be made based on the multidirectional model of functionality, which integrates the different dimensions, establishing relationships between the environment, the performance of activities and social participation.
Depression | Baseline and after 4 weeks
  The Beck Depression Inventory (BDI) - originally developed by Beck, Ward, Mendelson, Mock and Erbaugh (1961). It is a self-report scale to survey the intensity of depressive symptoms (Beck & Steer, 1993; Rosa, Malandrin, Leite & Silva, 1986), consisting of 21 items and reliability estimates established from six samples psychiatric disorders (Beck & Steer, 1993) that varied between 0.79 and 0.90.
Anxiety | Baseline and after 4 weeks
  State-Trait Anxiety Inventory (STAI) - It was prepared by Spielberger, Gorsuch and Lushene (1970) and translated and adapted to Brazil by Biaggio (Biaggio & Natalício 1979). Consisting of 2 self-report scales that assess anxiety as a state (STAI-E) or trait (STAI-T). Each situation (state and trait) has 20 items with scores from 1 to 4 in each one. The score ranges from 20 to 80. For each question the score corresponding to the answer is assigned, but for questions with a positive character the score is reversed.

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Principal Investigator — Federal University of Paraiba
Locations (1):
- Suellen Marinho Andrade, João Pessoa, Paraíba, Brazil

REFERENCES:
- [Derived] Ferreira CM, de Carvalho CD, Gomes R, Bonifacio de Assis ED, Andrade SM. Transcranial Direct Current Stimulation and Mirror Therapy for Neuropathic Pain After Brachial Plexus Avulsion: A Randomized, Double-Blind, Controlled Pilot Study. Front Neurol. 2020 Dec 11;11:568261. doi: 10.3389/fneur.2020.568261. eCollection 2020. PMID 33362687